CLINICAL TRIAL: NCT06539884
Title: Does the Phoenix Pediatric Sepsis Prognosis Prediction Scale Work
Status: Completed | Type: Observational
Sponsor: Oguz Dursun (Other)
Responsible Party: Sponsor-Investigator, Oguz Dursun, Prof. Dr., Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: TBAEK-391
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Sepsis; Sepsis, Severe
Keywords: Phoenix Score; 2005 SIRS (systemic inflammatory response syndrome); PRISM III (Pediatric Mortality Risk Score); PELOD II (Pediatric Logistic Organ Dysfunction); pSOFA (Pediatric sequential organ failure assessment)
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational — Evaluating whether the 2005 SIRS - Sepsis diagnostic and grading criteria, pSOFA, PRISM III and PELOD scores are compatible and to compare their prognostic predictive power.

SUMMARY:
The aim of this study to understand the compatibility of Phoenix Score, International 2005 SIRS criterias and PRISM III, PELOD scoring systems. Defining pediatric sepsis in our research, epidemiology, scoring systems and prognosis. In addition, we will evaluate the advantages and disadvantages of the Phoenix criteria and assess the compatibility in pediatric sepsis scoring systems. The subject of our research is the use of the Phoenix criteria for pediatric sepsis. The aim of this study was to evaluate whether the 2005 SIRS - Sepsis diagnostic and grading criteria, pSOFA, PRISM III and PELOD scores are compatible and to compare their prognostic predictive power. The study is a 1-year prospective observational study. Patients will not undergo any interventional procedure or blood tests due to this study. No intervention will be made in the treatment protocol.

In this study, Akdeniz University medical patients admitted to the Faculty of Pediatric Emergency Department with clinical sepsis suspicion will be included in the study. In 2024 it was aimed to evaluate whether the Phoenix criteria, which are recommended to be used to evaluate the prognosis of sepsis in pediatric patients, are compatible with the 2005 SIRS sepsis diagnosis and grading criteria, pSOFA, PRISM III and PELOD scores, which were widely used for this purpose in previous years and described in detail in the introduction section, and to compare their predictive power in terms of morbidity and mortality.

DETAILED DESCRIPTION:
Pediatric sepsis is a serious clinical syndrome leading to organ dysfunction develops in children due to infection. Various scoring systems are used to diagnose, treat and asses for pediatric sepsis. The most common of these Pediatric Risk of Mortality Score III (PRISM III) and Pediatric Logistic Organ Dysfunction (PELOD) scores. PRISM III is a set of 17 physiologic scores measured within the first 24 hours of ICU admission that predicts mortality risk based on the variable. In addition PELOD measures morbidity by assessing dysfunction in six organ systems. These scores are important in the management of pediatric sepsis.

tools, but they also have some limitations. For example, the PRISM III score, does not take into the reason for the admission, underlying disease, infectious agent and response to treatment of the patient. PELOD score does not reflect the duration and severity of organ dysfunction. Therefore, new studies and improvements in the definition of pediatric sepsis and scores are in progress. Pediatric SOFA (pSOFA) score is another option for definition and to approach the pediatric sepsis. It is used to assess the severity of sepsis and organ function in children. These criteria include respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. For each system, specific parameters are considered and scored. These scores are summed to calculate the SOFA score and the risk of organ failure is estimated. The Pediatric Functional Status Scale (FSS) is a rapid, objective and reliable tool used to assess the functional status of children during hospitalization. FSS, mental status, sensory function, communication, motor function, nutrition and respiratory status and each area is given a score between 1 (normal) and 5 (very severe dysfunction). Total scores range from 6 to 30. In recent years, a new set of criteria called the Phoenix criteria a definition of pediatric sepsis has been proposed. Phoenix criterias which includes both systemic inflammatory response syndrome (SIRS) and organ dysfunction criterias aims more accurate and early recognition of pediatric sepsis. Whether the Phoenix criteria are compatible with PRISM III and PELOD scores has not yet been investigated. The aim of this study to understand the compatibility of Phoenix Score, International 2005 SIRS criterias and PRISM III, PELOD scoring systems. Defining pediatric sepsis in our research, epidemiology, scoring systems and prognosis. In addition, we will evaluate the advantages and disadvantages of the Phoenix criteria and assess the compatibility in pediatric sepsis scoring systems. The subject of our research is the use of the Phoenix criteria for pediatric sepsis. The aim of this study was to evaluate whether the 2005 SIRS - Sepsis diagnostic and grading criteria, pSOFA, PRISM III and PELOD scores are compatible and to compare their prognostic predictive power. The study is a 1-year prospective observational study. Patients will not undergo any interventional procedure or blood tests due to this study. No intervention will be made in the treatment protocol.

In this study, Akdeniz University medical patients admitted to the Faculty of Pediatric Emergency Department with clinical sepsis suspicion will be included in the study. In 2024 it was aimed to evaluate whether the Phoenix criteria, which are recommended to be used to evaluate the prognosis of sepsis in pediatric patients, are compatible with the 2005 SIRS sepsis diagnosis and grading criteria, pSOFA, PRISM III and PELOD scores, which were widely used for this purpose in previous years and described in detail in the introduction section, and to compare their predictive power in terms of morbidity and mortality.

Patient/Volunteer/Participant definition and number: The patient group consisted of patients admitted to the Pediatric Emergency Department of Akdeniz University Faculty of Medicine who were clinically suspected of sepsis or admitted to the general pediatric service or pediatric intensive care unit with suspected sepsis. The study is a one-year prospective observational study. The number of patients will be determined by the number of patients admitted during this period and the group of patients with suspected sepsis.

ELIGIBILITY:
Inclusion criteria:

* Patients aged between 1 month to 18 years.
* Patients shall be suspected with sepsis clinically.

Exclusion criteria:

* Patients under 1 month of age.
* Patients over 18 years of age.
* Patients have not diagnostics of sepsis

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients aged 1 month to 18 years with clinically suspected sepsis will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Phoenix sepsis score correlates with length of stay in pediatric intensive care unit, length of stay in hospital, and mortality. | 1.5 year
  Phoenix sepsis score correlates with length of stay in pediatric intensive care unit, length of stay in hospital, and mortality.

SECONDARY OUTCOMES:
SOFA score correlates with length of stay in pediatric intensive care unit, length of stay in hospital, and mortality. | 1,5 year
  SOFA score correlates with length of stay in pediatric intensive care unit, length of stay in hospital, and mortality.
Phoenix sepsis score, SOFA score, and 2005 SIRS -sepsis definition define all children with sepsis. | 1,5 years
  Phoenix sepsis score, SOFA score, and 2005 SIRS -sepsis definition define all children with sepsis.
Phoenix sepsis score correlates with PRISM III, PELOD II scores, and the highest VIS observed during hospitalization. | 1,5 years
  Phoenix sepsis score correlates with PRISM III, PELOD II scores, and the highest VIS observed during hospitalization.
SOFA score correlates with PRISM III, PELOD II scores, and the highest VIS observed during hospitalization. | 1,5 years
  SOFA score correlates with PRISM III, PELOD II scores, and the highest VIS observed during hospitalization.
Phoenix sepsis score correlates with FSS calculated at discharge. | 1,5 years
  Phoenix sepsis score correlates with FSS calculated at discharge.
SOFA score correlates with FSS calculated at discharge. | 1,5 years
  SOFA score correlates with FSS calculated at discharge.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Akdeniz University, Antalya, Antalya
  - Akdeniz University, Konyaalti, Antalya

IPD SHARING:
Plan to Share IPD: No